CLINICAL TRIAL: NCT01399112
Title: A Usability Study of a Smoking Cessation Decision Aid in People With a Recent First Episode of Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Tara Mandel, Psychologist, Northwell Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EDSS
Record Dates: First submitted 2010-07-27; First posted 2011-07-21 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Smoking; Psychosis
Keywords: Smoking Cessation; First episode psychosis; Electronic Decision Support System
MeSH Terms: conditions — Smoking; Psychotic Disorders; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Decision Support System (Experimental): The Electronic Decision Support System (EDSS) is a 5-module computer program aimed to assess, motivate, educate, solicit preferences, and provide feedback and referrals for people with severe mental illness. The program provides: a) a personalized assessment of the individual's smoking, b) information to improve knowledge of smoking risks and treatment benefits, c) interactive exercises to personalize the impact of smoking, improve attitudes about quitting, and increase self-efficacy for seeking smoking cessation treatment, and d) a video patient vignette to develop social norms for smoking cessation treatment and increase self-efficacy. Usability testing among people with severe mental illness established that the system was comprehensible, easy to use, and took 30-90 minutes to complete.
  Interventions: Behavioral: Web-based computer program
- thetruth.com website (Active Comparator): Participants who are assigned to use the web-based thetruth.com website will be asked to navigate through the website as they wish. The home page of thetruth.com site has links to access video games, fact sheets, and videos that highlight negative aspects of cigarettes or tobacco companies. Thetruth.com website is not structured and participants can utilize whatever aspects of the website they wish and in any order they wish to view them.
  Individuals will use the computer with a research staff member present who can provide assistance if needed. The sections of the two programs website that are used and the time spend on each portion of the program will be recorded. Participants who use TheTruth.com will be given a referral for assistance in quitting smoking if requested.
  Interventions: Behavioral: Web-based computer program

INTERVENTIONS:
Behavioral: Web-based computer program — Web-based computer programs will be used to help education people with a recent first episode of a mental illness learn about smoking. The programs are designed to help young smokers become motivated to being a smoking cessation program.
  Other Names: EDSS

SUMMARY:
The investigators propose to recruit patients who have experienced a recent first episode of psychosis who have a chart diagnosis of Schizophrenia, Schizophrenifom, Schizoaffective Disorder, Psychosis NOS, or Bipolar I Disorder with psychotic features and self identify themselves as a current cigarette smoker. Aiding this population with smoking cessation is crucial as the majority of people with schizophrenia spectrum disorders (50-90%) smoke, which is leading to early mortality. While these individuals can benefit from standard evidence-based treatment, these treatments are underutilized. Web based programs, such as the EDSS and thetruth.com, can provide education and motivational tools to help people with a recent onset of psychosis use evidence-based smoking cessation treatments. This study aims to test these two web-based programs among young people with a recent episode of psychosis for usability and likeability and to explore whether use of these two programs will motivate users to seek smoking cessation treatment or to engage in other quitting behaviors in the month following use of the programs. Information gathered from this proposal will be used to help the researchers decide whether either of these two programs will be reasonable to include in a larger study of a comprehensive treatment for individuals with first episode psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnoses of Schizophrenia, Schizophrenifom, Schizoaffective Disorder, Psychosis NOS, or Bipolar I Disorder with psychotic features
* Diagnosed with one of above diagnoses within the past five years
* Ages 15-30 years old.
* Self-identified current cigarette smokers
* 5th grade reading level
* Willing to be audio recorded.
* Willing and legally able to provide informed consent to participate in the study or have a guardian provide informed consent with assent of a minor

Exclusion Criteria:

* Physically unable to use a computer with assistance.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
number of cigarettes smoked | One month
  Self-report of number of cigarettes smoked at baseline and at one month follow-up

SECONDARY OUTCOMES:
Satisfaction | Immediately (up to 10 minutes) following the use of one of the web-based programs.
  Immediately after using the assigned web-based program, the participant will be asked a series of questions regarding what they liked, did not like, found easy to use or found difficult to use when engaging with the computer program. These questions take approximately 5-10 minutes to answer.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Mandel, Ph.D., Principal Investigator — Northwell Health
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

REFERENCES:
- See also: thetruth.com website used as active comparison for EDSS — http://www.thetruth.com